CLINICAL TRIAL: NCT00822341
Title: A Randomized, Double-Blind, Placebo-Controlled, Sequential Ascending Single Intravenous Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TG-0054 in Healthy Subjects
Brief Title: Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of TG-0054 With Single IV Doses Escalation in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GPCR Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TG-0054-01
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: TG-0054 — 0.10, 0.14, 0.28, 0.56, 1.12, 2.24, 3.14, and 4.40 mg/kg of TG-0054/placebo via 15 min IV infusion

SUMMARY:
TG-0054 is a CXCR4 antagonist with stem cell mobilization effect as proven in animal model, this is the fist in human study to investigator the safety, tolerability and PK/PD in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female 18 to 45 years of age inclusive
* Body mass index (BMI) in the range of 19.0 to 30.0 kg/m² and body weight ≥ 50 kg inclusive
* Good physical and mental health status determined on the basis of the medical history and a general clinical examination
* Subjects must have used a consistent form of acceptable oral birth control or the double barrier method (intrauterine device (IUD) plus condom, spermicidal gel plus condom) for at least 3 months prior to study initiation

Exclusion Criteria:

* Any medical condition (other than a self-limited illness) that requires ongoing and current medical attention
* History of any other hematologic disorders including thromboembolic disease or anemia
* Severe trauma, fracture, major surgery, or biopsy of a parenchymal organ within the past 3 months
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent
* Subjects who currently smoke (intake nicotine or nicotine-containing products) or have given up smoking for less than 6 months before the first administration of study drug
* Subjects who are carriers of the Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody or who are Human Immunodeficiency Virus (HIV) antibody positive

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability for a single IV dose of TG-0054
To determine the maximum tolerated dose (MTD) of TG-0054

SECONDARY OUTCOMES:
To assess the plasma pharmacokinetics (PK) profile of TG-0054
To assess the pharmacodynamic (PD) effects of TG-0054 via CD34+stem cell, CD133+ progenitor cell counts; white blood cell (WBC), red blood cell (RBC), platelet, and differential counts

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, M.D., Principal Investigator — PAREXEL Clinical Pharmacology Research Unit Harbor Hospital Center
Locations (1):
- PAREXEL Clinical Pharmacology Research Unit Harbor Hospital Center, Baltimore, Maryland, United States